CLINICAL TRIAL: NCT00394108
Title: Changes in Cerebrovascular Reactivity During Cognitive Activation After Cardiopulmonary Bypass: Relation With Intraoperative Embolic Load and Postoperative Neuropsychological Dysfunctions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Fund for Scientific Research, Flanders, Belgium (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1997/098
Record Dates: First submitted 2006-10-30; First posted 2006-10-31 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: CABG-Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Determination of neuropsychological status

SUMMARY:
The study aims to evaluate neuropsychological disorders in CABG patients. Measurements are performed 1 day before, 6 days, 6 months and 3-5 years after the surgery. The relation with cerebrovascular reactivity and embolic load (measured by transcranial Doppler Ultrasonography) is evaluated. Two surgery techniques (on- and off-pump CABG) are compared.

ELIGIBILITY:
Inclusion Criteria:

* CABG-patients (not urgent)
* < 70 years old
* Righthanded

Exclusion Criteria:

* Neurological or psychiatric disease
* Psychoactive medication
* Valve operation

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 1999-08; Study Completion 2002-07 (Actual)

PRIMARY OUTCOMES:
Neuropsychological status | after 6 days, 6 months and 3-5 years

SECONDARY OUTCOMES:
Relation with intra-operative embolic load

CONTACTS AND LOCATIONS:
Overall Officials: Guy Vingerhoets, Psychologist, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be